CLINICAL TRIAL: NCT05335538
Title: The Role of TruGraf® to Optimize Outcomes in Pediatric Renal Transplantation
Brief Title: TruGraf and TRAC In Pediatrics Study
Acronym: TTIPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Transplant Genomics, Inc. (Industry)
Collaborators: University of Alabama at Birmingham (Other); University of British Columbia (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: TGRP08
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2021-08

CONDITIONS: Kidney Transplant Rejection
Keywords: Biomarkers; Subclinical Rejection; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Patients monitored with TruGraf and TRAC testing — This is an observational study there are no protocol mandated interventions. TruGraf and TRAC results will be utilized in conjunction with standard of care assessments to determine patient management.

SUMMARY:
This is a pilot 3 center prospective study of pediatric renal kidney recipients undergoing protocol biopsies examining the performance of the TruGraf gene expression test in children and adolescents.

DETAILED DESCRIPTION:
In pediatric renal transplant recipients, subclinical rejection in protocol biopsies is associated with a significantly increased incidence of acute rejection and/or allograft loss at 5 years post-transplant. Currently, TruGraf is the only noninvasive test designed and validated in adult kidney transplant recipients for use in ruling out silent subacute rejection in that has been approved by Medicare as an alternative to surveillance biopsies. The first step to the use of TruGraf in pediatrics is to perform a validation study in children and adolescents. Specifically, if validated in children and adolescents, a TruGraf result would enable a pediatric transplant physician to identify patients in whom no intervention is necessary without the need of a protocol biopsy. Therefore the aim of this study is to examine the concordance between the results of the TruGraf tests and protocol biopsies taken from stable pediatric renal transplant patients concurrently.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1-≤ 18 years and recipients of either living or deceased donor transplants Undergoing a protocol biopsy at either 3, 6, 12, 24 or 36 months
* Serum creatinine at the time of the clinic visit prior to the scheduled biopsy within 30% of a baseline calculated as the mean of the recipient's last 3 serum creatinine levels
* Serum creatinine level at the time of protocol biopsy ≤ 1.7 mg/dl.
* Patient receiving immunosuppression with a calcineurin inhibitor (either tacrolimus or cyclosporine) and/or an antimetabolite (either mycophenolate mofetil, mycophenolic acid EC or azathioprine) and/or an mTOR inhibitor (either sirolimus or everolimus) and/or corticosteroids.
* Absence of any systemic or urinary bacterial, viral or fungal infection
* Absence of significant BK viremia (as determined by the laboratory where the determination is run) at the time of the last clinical determination and at the time of the protocol biopsy
* Parents or guardians are capable of reading and understanding the Informed Consent document and willing to participate; if appropriate, patient is also able to understand the Informed Consent. If patient is older than 13 years, patient should be able to give Assent as written on Assent Form.
* For females of child-bearing age, a negative pregnancy test within 6 weeks of the protocol biopsy.

Exclusion Criteria:

* Refusal to undergo clinical standard-of-care protocol biopsy by either parent/guardian or patient.
* Inability to obtain adequate tissue on protocol biopsy
* Current participation in another interventional research study; patients who have completed the drug in another interventional study are eligible if they meet all other inclusion criteria.
* Serum creatinine at the clinic visit prior to the biopsy is > 30% of a baseline calculated as the mean of the recipient's last 3 serum creatinine levels.
* Serum creatinine at the time of the protocol biopsy ≥ 1.8 mg/dl. If the patient had a baseline < 1.8, and the creatinine on the day of biopsy is ≥ 1.8, at the discretion of the PI, the patient will be instructed to hydrate for 4 days and a serum creatinine will be obtained at that time. This is standard clinical practice. If the creatinine returns to the baseline (i.e., ≤ 30%) range, the patient will be classified as having stable renal function, while if the patient's serum creatinine does not return to the ≤ 30% range, he/she will be classified as having renal dysfunction
* Patients who, in the estimation of the investigator, are undergoing "for-cause" biopsies.
* Presence of any current and active bacterial, viral or fungal infection
* Presence of BK viremia judged to be significant by the site PI.
* Presence of BK nephropathy
* History of PTLD or malignancy
* Parents / guardians do not understand Informed Consent and / or are unwilling to participate; patient, if of appropriate age, is unwilling to participate
* Patients manifesting recurrent disease in their transplant (such as FSGS/nephrotic syndrome, C3 Glomeruopathy, MPGN, hyperoxaluria)
* Abnormal proteinuria as determined by a urinary protein: creatinine ratio of >1.
* Recipients of multi-organ transplants.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Renal transplant pediatric patients age 1 to 18 years old who must be undergoing a protocol biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Concordance of Biomarkers with protocol biopsy | 1 year
  Examination of the concordance between the results of the TruGraf tests and protocol biopsies taken from stable pediatric renal transplant concurrently.

SECONDARY OUTCOMES:
Concordance between the results of the TruGraf test and the histological finding of borderline changes vs. TCMR vs. AMR. | 1 year
  Separately examine the concordance between the results of the TruGraf test and the histological finding of borderline changes vs. TCMR vs. AMR.
Compare TruGraf results in patients ≤ 11 years old vs ≥ 12 years old | 1 year
  Compare the agreement between protocol biopsies and TruGraf results in patients ≤ 11 years old vs ≥ 12 years old
Relationship between de novo DSA, a normal protocol biopsy and the TruGraf result. | 1 year
  Assess the relationship, if any, between the appearance of de novo DSA, a normal protocol transplant biopsy and the TruGraf result.
Examine TruGraf results and the %CV tacrolimus levels- index of medication nonadherence. | 1 year
  Examine the relationship between the TruGraf results and the %CV tacrolimus levels as an index of medication nonadherence.
Relationship between urinary CXCL10 and subclinical rejection affecting the predictive value of TruGraf. | 1 year
  Examine the relationship between urinary CXCL10 and subclinical rejection in this patient cohort to examine whether it improves the performance metrics by improving the negative or positive predictive of TruGraf.
Examine relationship between ddcfDNA and subclinical rejection | 1 year
  Examine the relationship between ddcfDNA and subclinical rejection in this patient cohort

CONTACTS AND LOCATIONS:
Overall Officials: Patty West-Thielke, PharmD, Study Director — Transplant Genomics
Locations (3):
- United States (2):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA Mattel Children's Hospital, Los Angeles, California
- British Columbia Children's Hospital, Vancouver, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moudgil A, Dharnidharka VR, Lamb KE, Meier-Kriesche HU. Best allograft survival from share-35 kidney donors occurs in middle-aged adults and young children-an analysis of OPTN data. Transplantation. 2013 Jan 27;95(2):319-25. doi: 10.1097/TP.0b013e3182719203. PMID 23154211
- [Background] Horslen S, Barr ML, Christensen LL, Ettenger R, Magee JC. Pediatric transplantation in the United States, 1996-2005. Am J Transplant. 2007;7(5 Pt 2):1339-58. doi: 10.1111/j.1600-6143.2007.01780.x. PMID 17428284
- [Background] Verghese PS. Pediatric kidney transplantation: a historical review. Pediatr Res. 2017 Jan;81(1-2):259-264. doi: 10.1038/pr.2016.207. Epub 2016 Oct 12. PMID 27732587
- [Background] United States Renal Data System 2018 Annual Data Report Volume 2 ESRD Chapter 5
- [Background] Aubert O, Loupy A, Hidalgo L, Duong van Huyen JP, Higgins S, Viglietti D, Jouven X, Glotz D, Legendre C, Lefaucheur C, Halloran PF. Antibody-Mediated Rejection Due to Preexisting versus De Novo Donor-Specific Antibodies in Kidney Allograft Recipients. J Am Soc Nephrol. 2017 Jun;28(6):1912-1923. doi: 10.1681/ASN.2016070797. Epub 2017 Mar 2. PMID 28255002
- [Background] Ettenger R, Albrecht R, Alloway R, Belen O, Cavaille-Coll MW, Chisholm-Burns MA, Dew MA, Fitzsimmons WE, Nickerson P, Thompson G, Vaidya P. Meeting report: FDA public meeting on patient-focused drug development and medication adherence in solid organ transplant patients. Am J Transplant. 2018 Mar;18(3):564-573. doi: 10.1111/ajt.14635. Epub 2018 Jan 25. PMID 29288623
- [Background] Birk PE. Surveillance biopsies in children post-kidney transplant. Pediatr Nephrol. 2012 May;27(5):753-60. doi: 10.1007/s00467-011-1969-8. Epub 2011 Jul 27. PMID 21792611
- [Background] Gordillo R, Munshi R, Monroe EJ, Shivaram GM, Smith JM. Benefits and risks of protocol biopsies in pediatric renal transplantation. Pediatr Nephrol. 2019 Apr;34(4):593-598. doi: 10.1007/s00467-018-3959-6. Epub 2018 May 3. PMID 29725772
- [Background] Nazario M, Nicoara O, Becton L, Self S, Hill J, Mack E, Evans M, Twombley K. Safety and utility of surveillance biopsies in pediatric kidney transplant patients. Pediatr Transplant. 2018 Jun;22(4):e13178. doi: 10.1111/petr.13178. Epub 2018 Mar 27. PMID 29582530
- [Background] Rush D. Protocol biopsies should be part of the routine management of kidney transplant recipients. Pro. Am J Kidney Dis. 2002 Oct;40(4):671-3. doi: 10.1053/ajkd.2002.36427. No abstract available. PMID 12324898
- [Background] Rose EM, Kennedy SE, Mackie FE. Surveillance biopsies after paediatric kidney transplantation: A review. Pediatr Transplant. 2016 Sep;20(6):748-55. doi: 10.1111/petr.12733. Epub 2016 Jun 16. PMID 27306873
- [Background] Birk PE, Stannard KM, Konrad HB, Blydt-Hansen TD, Ogborn MR, Cheang MS, Gartner JG, Gibson IW. Surveillance biopsies are superior to functional studies for the diagnosis of acute and chronic renal allograft pathology in children. Pediatr Transplant. 2004 Feb;8(1):29-38. doi: 10.1046/j.1397-3142.2003.00122.x. PMID 15009838
- [Background] Furness PN, Philpott CM, Chorbadjian MT, Nicholson ML, Bosmans JL, Corthouts BL, Bogers JJ, Schwarz A, Gwinner W, Haller H, Mengel M, Seron D, Moreso F, Canas C. Protocol biopsy of the stable renal transplant: a multicenter study of methods and complication rates. Transplantation. 2003 Sep 27;76(6):969-73. doi: 10.1097/01.TP.0000082542.99416.11. PMID 14508363
- [Background] Nankivell BJ, Agrawal N, Sharma A, Taverniti A, P'Ng CH, Shingde M, Wong G, Chapman JR. The clinical and pathological significance of borderline T cell-mediated rejection. Am J Transplant. 2019 May;19(5):1452-1463. doi: 10.1111/ajt.15197. Epub 2019 Jan 22. PMID 30501008
- [Background] Seifert ME, Yanik MV, Feig DI, Hauptfeld-Dolejsek V, Mroczek-Musulman EC, Kelly DR, Rosenblum F, Mannon RB. Subclinical inflammation phenotypes and long-term outcomes after pediatric kidney transplantation. Am J Transplant. 2018 Sep;18(9):2189-2199. doi: 10.1111/ajt.14933. Epub 2018 Jun 27. PMID 29766640
- [Background] Loupy A, Vernerey D, Tinel C, Aubert O, Duong van Huyen JP, Rabant M, Verine J, Nochy D, Empana JP, Martinez F, Glotz D, Jouven X, Legendre C, Lefaucheur C. Subclinical Rejection Phenotypes at 1 Year Post-Transplant and Outcome of Kidney Allografts. J Am Soc Nephrol. 2015 Jul;26(7):1721-31. doi: 10.1681/ASN.2014040399. Epub 2015 Jan 2. PMID 25556173
- [Background] Beimler J, Zeier M. Borderline rejection after renal transplantation--to treat or not to treat. Clin Transplant. 2009 Dec;23 Suppl 21:19-25. doi: 10.1111/j.1399-0012.2009.01105.x. PMID 19930312
- [Background] Bunchman TE, Fryd DS, Sibley RK, Mauer SM. Manifestations of renal allograft rejection in small children receiving adult kidneys. Pediatr Nephrol. 1990 May;4(3):255-8. doi: 10.1007/BF00857670. PMID 2400654
- [Background] Foster BJ, Dahhou M, Zhang X, Platt RW, Samuel SM, Hanley JA. Association between age and graft failure rates in young kidney transplant recipients. Transplantation. 2011 Dec 15;92(11):1237-43. doi: 10.1097/TP.0b013e31823411d7. PMID 22124283
- [Background] Ettenger RB, Tsai EW, Fine RN. A paradigm shift and a few modest suggestions in the care of adolescent transplant recipients. Transplantation. 2011 Dec 15;92(11):1191-3. doi: 10.1097/TP.0b013e318238da81. No abstract available. PMID 22081055
- [Background] Pizzo HP, Ettenger RB, Gjertson DW, Reed EF, Zhang J, Gritsch HA, Tsai EW. Sirolimus and tacrolimus coefficient of variation is associated with rejection, donor-specific antibodies, and nonadherence. Pediatr Nephrol. 2016 Dec;31(12):2345-2352. doi: 10.1007/s00467-016-3422-5. Epub 2016 Jun 10. PMID 27286686
- [Background] Parajuli S, Reville PK, Ellis TM, Djamali A, Mandelbrot DA. Utility of protocol kidney biopsies for de novo donor-specific antibodies. Am J Transplant. 2017 Dec;17(12):3210-3218. doi: 10.1111/ajt.14466. Epub 2017 Sep 26. PMID 28805293
- [Background] Robert Ettenger and Margaret L. Stuber. Nonadherence, Psychosocial Adaptation and Its Effects in Pediatric Transplantation. In Textbook of Organ Transplantation, First Edition. Edited by Allan D. Kirk, Stuart J. Knechtle, Christian P. Larsen, Joren C. Madsen, Thomas C. Pearson, and Steven A. Webber. © 2014 John Wiley & Sons, Ltd. Published 2014 by John Wiley & Sons, Ltd.
- [Background] Hsiau M, Fernandez HE, Gjertson D, Ettenger RB, Tsai EW. Monitoring nonadherence and acute rejection with variation in blood immunosuppressant levels in pediatric renal transplantation. Transplantation. 2011 Oct 27;92(8):918-22. doi: 10.1097/TP.0b013e31822dc34f. PMID 21857278
- [Background] Benfield MR, Herrin J, Feld L, Rose S, Stablein D, Tejani A. Safety of kidney biopsy in pediatric transplantation: a report of the Controlled Clinical Trials in Pediatric Transplantation Trial of Induction Therapy Study Group. Transplantation. 1999 Feb 27;67(4):544-7. doi: 10.1097/00007890-199902270-00010. PMID 10071025
- [Background] Thaunat O, Legendre C, Morelon E, Kreis H, Mamzer-Bruneel MF. To biopsy or not to biopsy? Should we screen the histology of stable renal grafts? Transplantation. 2007 Sep 27;84(6):671-6. doi: 10.1097/01.tp.0000282870.71282.ed. PMID 17893596
- [Background] Dharnidharka VR, Malone A. Biomarkers to detect rejection after kidney transplantation. Pediatr Nephrol. 2018 Jul;33(7):1113-1122. doi: 10.1007/s00467-017-3712-6. Epub 2017 Jun 19. PMID 28631040
- [Background] Naesens M, Friedewald J, Mas V, Kaplan B, Abecassis MM. A Practical Guide to the Clinical Implementation of Biomarkers for Subclinical Rejection Following Kidney Transplantation. Transplantation. 2020 Apr;104(4):700-707. doi: 10.1097/TP.0000000000003064. PMID 31815910
- [Background] Wiebe C, Nickerson P. Posttransplant monitoring of de novo human leukocyte antigen donor-specific antibodies in kidney transplantation. Curr Opin Organ Transplant. 2013 Aug;18(4):470-7. doi: 10.1097/MOT.0b013e3283626149. PMID 23695596
- [Background] Wu P, Everly MJ, Rebellato LM, Haisch CE, Briley KP, Bolin P, Kendrick WT, Kendrick SA, Morgan C, Harland RC, Terasaki PI. Trends and characteristics in early glomerular filtration rate decline after posttransplantation alloantibody appearance. Transplantation. 2013 Nov 27;96(10):919-25. doi: 10.1097/TP.0b013e3182a289ac. PMID 23912173
- [Background] Engen RM, Park GE, Schumacher CS, Gimferrer I, Warner P, Finn LS, Weiss NS, Smith JM. Donor-specific Antibody Surveillance and Graft Outcomes in Pediatric Kidney Transplant Recipients. Transplantation. 2018 Dec;102(12):2072-2079. doi: 10.1097/TP.0000000000002310. PMID 29863579
- [Background] Roedder S, Sigdel T, Salomonis N, Hsieh S, Dai H, Bestard O, Metes D, Zeevi A, Gritsch A, Cheeseman J, Macedo C, Peddy R, Medeiros M, Vincenti F, Asher N, Salvatierra O, Shapiro R, Kirk A, Reed EF, Sarwal MM. The kSORT assay to detect renal transplant patients at high risk for acute rejection: results of the multicenter AART study. PLoS Med. 2014 Nov 11;11(11):e1001759. doi: 10.1371/journal.pmed.1001759. eCollection 2014 Nov. PMID 25386950
- [Background] Rush DN, Gibson IW. Subclinical Inflammation in Renal Transplantation. Transplantation. 2019 Jun;103(6):e139-e145. doi: 10.1097/TP.0000000000002682. PMID 30801537
- [Background] Kurian SM, Williams AN, Gelbart T, Campbell D, Mondala TS, Head SR, Horvath S, Gaber L, Thompson R, Whisenant T, Lin W, Langfelder P, Robison EH, Schaffer RL, Fisher JS, Friedewald J, Flechner SM, Chan LK, Wiseman AC, Shidban H, Mendez R, Heilman R, Abecassis MM, Marsh CL, Salomon DR. Molecular classifiers for acute kidney transplant rejection in peripheral blood by whole genome gene expression profiling. Am J Transplant. 2014 May;14(5):1164-72. doi: 10.1111/ajt.12671. Epub 2014 Apr 11. PMID 24725967
- [Background] Blydt-Hansen TD, Gibson IW, Gao A, Dufault B, Ho J. Elevated urinary CXCL10-to-creatinine ratio is associated with subclinical and clinical rejection in pediatric renal transplantation. Transplantation. 2015 Apr;99(4):797-804. doi: 10.1097/TP.0000000000000419. PMID 25222013
- [Background] Mockler C, Sharma A, Gibson IW, Gao A, Wong A, Ho J, Blydt-Hansen TD. The prognostic value of urinary chemokines at 6 months after pediatric kidney transplantation. Pediatr Transplant. 2018 Aug;22(5):e13205. doi: 10.1111/petr.13205. Epub 2018 May 7. PMID 29733487
- [Background] Matz M, Beyer J, Wunsch D, Mashreghi MF, Seiler M, Pratschke J, Babel N, Volk HD, Reinke P, Kotsch K. Early post-transplant urinary IP-10 expression after kidney transplantation is predictive of short- and long-term graft function. Kidney Int. 2006 May;69(9):1683-90. doi: 10.1038/sj.ki.5000343. PMID 16572110
- [Background] Tatapudi RR, Muthukumar T, Dadhania D, Ding R, Li B, Sharma VK, Lozada-Pastorio E, Seetharamu N, Hartono C, Serur D, Seshan SV, Kapur S, Hancock WW, Suthanthiran M. Noninvasive detection of renal allograft inflammation by measurements of mRNA for IP-10 and CXCR3 in urine. Kidney Int. 2004 Jun;65(6):2390-7. doi: 10.1111/j.1523-1755.2004.00663.x. PMID 15149352
- [Background] Hricik DE, Nickerson P, Formica RN, Poggio ED, Rush D, Newell KA, Goebel J, Gibson IW, Fairchild RL, Riggs M, Spain K, Ikle D, Bridges ND, Heeger PS; CTOT-01 consortium. Multicenter validation of urinary CXCL9 as a risk-stratifying biomarker for kidney transplant injury. Am J Transplant. 2013 Oct;13(10):2634-44. doi: 10.1111/ajt.12426. Epub 2013 Aug 22. PMID 23968332
- [Background] Bloom RD, Bromberg JS, Poggio ED, Bunnapradist S, Langone AJ, Sood P, Matas AJ, Mehta S, Mannon RB, Sharfuddin A, Fischbach B, Narayanan M, Jordan SC, Cohen D, Weir MR, Hiller D, Prasad P, Woodward RN, Grskovic M, Sninsky JJ, Yee JP, Brennan DC; Circulating Donor-Derived Cell-Free DNA in Blood for Diagnosing Active Rejection in Kidney Transplant Recipients (DART) Study Investigators. Cell-Free DNA and Active Rejection in Kidney Allografts. J Am Soc Nephrol. 2017 Jul;28(7):2221-2232. doi: 10.1681/ASN.2016091034. Epub 2017 Mar 9. PMID 28280140
- [Background] Huang E, Sethi S, Peng A, Najjar R, Mirocha J, Haas M, Vo A, Jordan SC. Early clinical experience using donor-derived cell-free DNA to detect rejection in kidney transplant recipients. Am J Transplant. 2019 Jun;19(6):1663-1670. doi: 10.1111/ajt.15289. Epub 2019 Mar 29. PMID 30725531
- [Background] Naesens M, Anglicheau D. Precision Transplant Medicine: Biomarkers to the Rescue. J Am Soc Nephrol. 2018 Jan;29(1):24-34. doi: 10.1681/ASN.2017010004. Epub 2017 Oct 9. PMID 28993504
- [Background] Anglicheau D, Naesens M, Essig M, Gwinner W, Marquet P. Establishing Biomarkers in Transplant Medicine: A Critical Review of Current Approaches. Transplantation. 2016 Oct;100(10):2024-38. doi: 10.1097/TP.0000000000001321. PMID 27479159
- [Background] Suthanthiran M, Schwartz JE, Ding R, Abecassis M, Dadhania D, Samstein B, Knechtle SJ, Friedewald J, Becker YT, Sharma VK, Williams NM, Chang CS, Hoang C, Muthukumar T, August P, Keslar KS, Fairchild RL, Hricik DE, Heeger PS, Han L, Liu J, Riggs M, Ikle DN, Bridges ND, Shaked A; Clinical Trials in Organ Transplantation 04 (CTOT-04) Study Investigators. Urinary-cell mRNA profile and acute cellular rejection in kidney allografts. N Engl J Med. 2013 Jul 4;369(1):20-31. doi: 10.1056/NEJMoa1215555. PMID 23822777
- [Background] Lo DJ, Kaplan B, Kirk AD. Biomarkers for kidney transplant rejection. Nat Rev Nephrol. 2014 Apr;10(4):215-25. doi: 10.1038/nrneph.2013.281. Epub 2014 Jan 21. PMID 24445740
- [Background] Abecassis M, Kaplan B. Transplantation: Biomarkers in transplantation-the devil is in the detail. Nat Rev Nephrol. 2015 Apr;11(4):204-5. doi: 10.1038/nrneph.2015.2. Epub 2015 Jan 27. No abstract available. PMID 25623476
- [Background] Peddi VR, Patel PS, Schieve C, Rose S, First MR. Serial Peripheral Blood Gene Expression Profiling to Assess Immune Quiescence in Kidney Transplant Recipients with Stable Renal Function. Ann Transplant. 2020 Apr 28;25:e920839. doi: 10.12659/AOT.920839. PMID 32341330
- [Background] Friedewald JJ, Kurian SM, Heilman RL, Whisenant TC, Poggio ED, Marsh C, Baliga P, Odim J, Brown MM, Ikle DN, Armstrong BD, Charette JI, Brietigam SS, Sustento-Reodica N, Zhao L, Kandpal M, Salomon DR, Abecassis MM; Clinical Trials in Organ Transplantation 08 (CTOT-08). Development and clinical validity of a novel blood-based molecular biomarker for subclinical acute rejection following kidney transplant. Am J Transplant. 2019 Jan;19(1):98-109. doi: 10.1111/ajt.15011. Epub 2018 Aug 31. PMID 29985559
- [Background] Mehta R, Cherikh W, Sood P, Hariharan S. Kidney allograft surveillance biopsy practices across US transplant centers: A UNOS survey. Clin Transplant. 2017 May;31(5). doi: 10.1111/ctr.12945. Epub 2017 Mar 23. PMID 28251702
- [Background] First MR, Peddi VR, Mannon R, Knight R, Marsh CL, Kurian SM, Rice JC, Maluf D, Mandelbrot D, Patel A, David J, Schieve C, Lee D, Lewis P, Friedewald JJ, Abecassis MM, Rose S. Investigator Assessment of the Utility of the TruGraf Molecular Diagnostic Test in Clinical Practice. Transplant Proc. 2019 Apr;51(3):729-733. doi: 10.1016/j.transproceed.2018.10.024. Epub 2018 Dec 11. PMID 30979457
- [Background] Marsh CL, Kurian SM, Rice JC, Whisenant TC, David J, Rose S, Schieve C, Lee D, Case J, Barrick B, Peddi VR, Mannon RB, Knight R, Maluf D, Mandelbrot D, Patel A, Friedewald JJ, Abecassis MM, First MR. Application of TruGraf v1: A Novel Molecular Biomarker for Managing Kidney Transplant Recipients With Stable Renal Function. Transplant Proc. 2019 Apr;51(3):722-728. doi: 10.1016/j.transproceed.2019.01.054. Epub 2019 Jan 26. PMID 30979456
- [Background] Naesens M. The special relativity of noninvasive biomarkers for acute rejection. Am J Transplant. 2019 Jan;19(1):5-8. doi: 10.1111/ajt.15078. Epub 2018 Sep 17. No abstract available. PMID 30125470
- [Background] Friedewald J, Abecassis M. Clinical implications for the use of a biomarker for subclinical rejection - Conflating arguments cause a disconnection between the premise and the conclusion. Am J Transplant. 2019 Jul;19(7):2141-2142. doi: 10.1111/ajt.15327. Epub 2019 Mar 18. No abstract available. PMID 30809931
- [Background] First MR, Whisenant T, Friedewald JJ, Lewis P, Rose S, et al. (2017) Clinical Utility of Peripheral Blood Gene Expression Profiling of Kidney Transplant Recipients to Assess the Need for Surveillance Biopsies in Subjects with Stable Renal Function. J Transplant Technol Res 7: 177.
- [Background] Loupy A, Haas M, Roufosse C, Naesens M, Adam B, Afrouzian M, Akalin E, Alachkar N, Bagnasco S, Becker JU, Cornell LD, Clahsen-van Groningen MC, Demetris AJ, Dragun D, Duong van Huyen JP, Farris AB, Fogo AB, Gibson IW, Glotz D, Gueguen J, Kikic Z, Kozakowski N, Kraus E, Lefaucheur C, Liapis H, Mannon RB, Montgomery RA, Nankivell BJ, Nickeleit V, Nickerson P, Rabant M, Racusen L, Randhawa P, Robin B, Rosales IA, Sapir-Pichhadze R, Schinstock CA, Seron D, Singh HK, Smith RN, Stegall MD, Zeevi A, Solez K, Colvin RB, Mengel M. The Banff 2019 Kidney Meeting Report (I): Updates on and clarification of criteria for T cell- and antibody-mediated rejection. Am J Transplant. 2020 Sep;20(9):2318-2331. doi: 10.1111/ajt.15898. Epub 2020 May 28. PMID 32463180
- [Background] Schaub S, Nickerson P, Rush D, Mayr M, Hess C, Golian M, Stefura W, Hayglass K. Urinary CXCL9 and CXCL10 levels correlate with the extent of subclinical tubulitis. Am J Transplant. 2009 Jun;9(6):1347-53. doi: 10.1111/j.1600-6143.2009.02645.x. Epub 2009 May 13. PMID 19459809
- [Background] Ho J, Rush DN, Karpinski M, Storsley L, Gibson IW, Bestland J, Gao A, Stefura W, HayGlass KT, Nickerson PW. Validation of urinary CXCL10 as a marker of borderline, subclinical, and clinical tubulitis. Transplantation. 2011 Oct 27;92(8):878-82. doi: 10.1097/TP.0b013e31822d4de1. PMID 21876477
- [Background] Rodrigo E, Segundo DS, Fernandez-Fresnedo G, Lopez-Hoyos M, Benito A, Ruiz JC, de Cos MA, Arias M. Within-Patient Variability in Tacrolimus Blood Levels Predicts Kidney Graft Loss and Donor-Specific Antibody Development. Transplantation. 2016 Nov;100(11):2479-2485. doi: 10.1097/TP.0000000000001040. PMID 26703349
- [Background] Kurian SM, Velazquez E, Thompson R, Whisenant T, Rose S, Riley N, Harrison F, Gelbart T, Friedewald JJ, Charette J, Brietigam S, Peysakhovich J, First MR, Abecassis MM, Salomon DR. Orthogonal Comparison of Molecular Signatures of Kidney Transplants With Subclinical and Clinical Acute Rejection: Equivalent Performance Is Agnostic to Both Technology and Platform. Am J Transplant. 2017 Aug;17(8):2103-2116. doi: 10.1111/ajt.14224. Epub 2017 Apr 3. PMID 28188669
- [Background] Ang A, Schieve C, Rose S, Kew C, First MR, Mannon RB. Avoiding surveillance biopsy: Use of a noninvasive biomarker assay in a real-life scenario. Clin Transplant. 2021 Jan;35(1):e14145. doi: 10.1111/ctr.14145. Epub 2020 Nov 24. PMID 33170974
- [Background] Li J, Fine J. On sample size for sensitivity and specificity in prospective diagnostic accuracy studies. Stat Med. 2004 Aug 30;23(16):2537-50. doi: 10.1002/sim.1836. PMID 15287083
- [Background] Kanzelmeyer NK, Ahlenstiel T, Drube J, Froede K, Kreuzer M, Broecker V, Ehrich JH, Melk A, Pape L. Protocol biopsy-driven interventions after pediatric renal transplantation. Pediatr Transplant. 2010 Dec;14(8):1012-8. doi: 10.1111/j.1399-3046.2010.01399.x. Epub 2010 Sep 15. PMID 20846241